CLINICAL TRIAL: NCT05264194
Title: The Effect of Continuous Versus Interrupted Suturing Technique on Perineal Pain After Perineorrhaphy: A Randomized Controlled Pilot Study
Brief Title: Suturing Techniques on Perineal Pain
Acronym: PNO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 12411
Record Dates: First submitted 2022-01-26; First posted 2022-03-03 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Perineal Pain
MeSH Terms: interventions — Suture Techniques

STUDY DESIGN:
Intervention Model Description: Patients will be randomly assigned to receive sutures that will either be hidden underneath their skin (subcuticular) or on your skin (transcutaneous) at the time of skin closure post-surgery.
Masking Description: Given the nature of the suturing techniques, it would be impossible to blind the study to the investigators and the participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients receiving subcuticular suturing (Active Comparator): Sutures will be hidden underneath skin
  Interventions: Other: Suturing technique
- Patients receiving transcutaneous suturing (Active Comparator): Sutures will be on your skin
  Interventions: Other: Suturing technique

INTERVENTIONS:
Other: Suturing technique — The technique (subcuticular or transcutaneous) that will be used to close skin post-surgery.

SUMMARY:
Perineorrhaphy, sometimes referred to as perineoplasty, is a common procedure in pelvic reconstructive surgery that entails surgical repair of the perineum. Indications may include: prevention of recurrent prolapse, treatment of pain, and improved sexual function and cosmesis, as well as to treat the sensation of a "wide vagina." Differences in postoperative pain by suturing technique and standard use of suture type are not well established. Patient satisfaction can be influenced by patient perceptions regarding postoperative pain, therefore reducing postoperative pain scores remains a priority. It is unclear whether suturing technique is associated with less pain after this procedure. Based on studies on repair of obstetric lacerations, we hypothesize that a subcuticular skin closure will be associated with less postoperative perineal pain compared to interrupted transcutaneous sutures.

DETAILED DESCRIPTION:
Recruitment will be carried out at OU Medical Center within a 12-month period either at OU Women's Pelvic and Bladder Health Clinic or OU Women's Health Clinic. Women who are planning pelvic organ prolapse repair and who are found to have genital hiatus of ≥4 cm on the pelvic organ prolapse quantification exam will be approached for study inclusion. A 4-cm or greater dimension of genital hiatus is associated with greater risk of prolapse recurrence, and researchers anticipate patients with this measurement prior to surgery will require a perineorrhaphy. These surgeries will be performed by one of two board certified female pelvic medicine and reconstructive surgery specialists. Given the nature of the suturing techniques, it would be impossible to blind the study to both the investigators and the participants.

Randomization will be completed prior to the procedure and contained within opaque sealed envelopes until a decision is made to proceed with a perineorrhaphy intraoperatively.

To standardize the procedure, an instructional video will be made to describe the subcuticular and transcutaneous interrupted techniques. This will serve as reference for investigators to adhere to the standard procedure. An educational webinar will be performed at the onset of the study and this instructional video will be available for review at any additional point during the study. Participants will be asked to complete a baseline SPS questionnaire prior to surgery. Perineorrhaphy will be carried out in our standard fashion and finalized with interrupted stitches of delayed absorbable monofilament sutures for reconstruction of the perineal body. The perineal skin closure will be randomized to continuous subcuticular or interrupted transcutaneous stitches of 3-0 polyglactin-910 (Vicryl). Researchers will follow the standard Enhanced Recovery After Anesthesia (ERAS) protocol for postoperative oral analgesia. Participants will be asked to complete daily SPS questionnaires in the first two weeks postoperatively. Patients are routinely scheduled for a 2- week and 3- month postoperative visit. Participants will complete a questionnaire to assess pain (SPS) and patient satisfaction at both visits. A pelvic exam is not routinely performed at the 2-week visit unless indicated otherwise by patient or provider concerns. At the 3-month postoperative visit, a sexual function questionnaire and a pelvic exam will be completed in addition to the pain and patient satisfaction survey. These surveys can be administered in person or remotely (by telephone or virtually), depending on the nature of the postoperative visits.

ELIGIBILITY:
Inclusion Criteria:

1. Women 18 years or greater planning pelvic floor surgery reconstruction
2. Genital hiatus on POP-Q exam of ≥4 cm

Exclusion Criteria:

1. History of pelvic radiation
2. History of chronic perineal pain or pudendal neuralgia
3. Planning on having an obliterative vaginal procedure.
4. Concomitant hemorrhoidectomy or colorectal procedure
5. Concomitant mesh removal procedure
6. Allergy to polyglycolic acid sutures
7. History of connective tissue disorder.
8. Chronic immunosuppression

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This study involves those undergoing a pelvic reconstructive surgery, more common for women.
Enrollment: 102 (Actual)
Dates: Start 2020-10-10 (Actual); Primary Completion 2023-01-09 (Actual); Study Completion 2023-01-09 (Actual)

PRIMARY OUTCOMES:
Pain level | 2 weeks
  Participants will complete a Situational Pain Scale (SPS) questionnaire. Pain on the SPS is measured from 0 (no pain sensation) to 10 (most intense pain imaginable).

SECONDARY OUTCOMES:
Patient satisfaction | 2 weeks
  Measured using a questionnaire from 1 (very unsatisfied) to 5 (very satisfied).
Perineal pain complications | 3 months
  Measured using pelvic exam.
Perineal pain complications | 3 months
  Measured using patient complaints.

CONTACTS AND LOCATIONS:
Overall Officials: Lieschen Quiroz, MD, Principal Investigator — University of Oklahoma HSC
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States